CLINICAL TRIAL: NCT01779466
Title: A Double-blind, Randomised, Parallel-group Trial Investigating Sleep Behaviour and Daytime Performance in Nocturia Patients Treated With Desmopressin Orally Disintegrating Tablets as Compared to Placebo
Brief Title: Daytime Impact Sleep Study
Acronym: DAISS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of eligible patients
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000088; 2012-004388-34 (EudraCT Number)
Record Dates: First submitted 2013-01-23; First posted 2013-01-30 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental A (Experimental)
  Interventions: Drug: Desmopressin
- Experimental B (Experimental)
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (not active)

INTERVENTIONS:
Drug: Desmopressin
  Arms: Experimental A; Experimental B
Drug: Placebo (not active)
  Arms: Placebo

SUMMARY:
This trial will investigate the relationship of sleep, daytime performance and nocturia in patients treated with Desmopressin or placebo. Male and Female patients will be administered Desmopressin or Placebo every day for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 night time voids per night
* Habitual sleep of 6-9.5 hours per night
* Experiencing symptoms of Nocturia greater than 6 months

Exclusion Criteria:

* Greater than 10 night time voids
* History of sleep apnoea and PLMS (Periodic Limb Movements of Sleep)
* Other sleep disorders
* Signs or symptoms of: Bladder outlet obstruction, severe lower urinary tract symptoms (LUTS), interstitial cystitis, moderate to severe overactive bladder (OAB), moderate to severe as judged by the investigator stress urinary incontinence
* Urological malignancies
* Neurogenic detrusor over activity (e.g. Parkinson, spinal cord damage, etc.)
* Central or nephrogenic diabetes insipidus
* Habitual or psychogenic polydipsia (fluid intake resulting in a urine production exceeding 40ml/Kg/24hrs)
* Syndrome of inappropriate antidiuretic hormone (SIADH)
* Cardiac failure evidence based on physical examination, cardiac medical history and electrocardiogram (ECG) output
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Hyponatraemia with sodium <135 mmol/L
* Renal insufficiency
* Known or suspected clinically significant hepatic and/or biliary diseases

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean number of nocturnal voids | 1 month and 3 months
  As measured by voiding diary
Wake after sleep onset | 1 month and 3 months
  i.e. time in minutes of epochs scored as wake from sleep onset latency until lights on. Measured by Polysomnography
Daytime sleepiness score as measured by Karolinska Sleepiness Scale and Epworth Sleepiness Scale | 1 month and 3 months
  Daytime performance
Mean time to first void | 1 month and 3 months
  As measured by voiding diary
Sleep efficiency | 1 month and 3 months
  Sleep efficiency equals total sleep time divided by total recording time multiplied by 100. Measured by Polysomnography
Sleep stage N1, N2, N3, (sleep stages in NREM (non-rapid eye movement) and REM (rapid eye movement) as a percentage of total sleep time | 1 month and 3 months
  Measured by Polysomnography
Number of awakenings due to nocturia | 1 month and 3 months
  Measured by Polysomnography
Latency to slow-wave sleep | 1 month and 3 months
  Measured by Polysomnography
Wake after sleep onset (WASO) i.e total minutes of wakefulness recorded after sleep onset | 1 month and 3 months
  Measured by Actigraphy
Percent of sleep | 1 month and 3 months
  Measured by Actigraphy
Number of awakenings due to nocturia | 1 month and 3 months
  Measured by Actigraphy
Quality of life score measured by EQ-5D-5L | 1 month and 3 months
  Daytime performance
Safety - incidence of adverse events | 1 month and 3 months
Safety - clinically significant changes in lab values | 1 week and 3 months
Safety - clinically significant changes in vital signs | 1 week, 1 month and 3 months
Safety - clinically significant changes in physical examination | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Surrey Clinical Research Centre, Surrey, United Kingdom